CLINICAL TRIAL: NCT02277652
Title: Comparison of Four Different Endotracheal Intubation Devices Performed by Emergency Medical Professionals: a Manikin Study With 6 Airway Scenarios
Brief Title: Endotracheal Intubation Devices
Acronym: ETID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ETI/2014/03
Record Dates: First submitted 2014-10-26; First posted 2014-10-29 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Scenario 1: Uninterrupted chest compressions (Experimental): Endotracheal intubation (ETI) during pediatric manikin with uninterrupted chest compressions. Chest compression was performed using LUCAS-2 (Physio-Control, USA).
  Interventions: Device: The Miller Laryngoscope; Device: The Bonfils intubation fibrescope; Device: The GlideScope Ranger; Device: The Supraglottic Airway Laryngopharyngeal Tube (SALT)
- Scenario 2: Neutral position (Experimental): ETI performed in neutral mannikin head position
  Interventions: Device: The Miller Laryngoscope; Device: The Bonfils intubation fibrescope; Device: The GlideScope Ranger; Device: The Supraglottic Airway Laryngopharyngeal Tube (SALT)
- Scenario 3: Sniffing position (Experimental): ETI performed in sniffing mannikin head position
  Interventions: Device: The Miller Laryngoscope; Device: The Bonfils intubation fibrescope; Device: The GlideScope Ranger; Device: The Supraglottic Airway Laryngopharyngeal Tube (SALT)
- Scenario 4: Pharyngeal swelling (Experimental): ETI performed during mannikin pharyngeal swelling scenario
  Interventions: Device: The Miller Laryngoscope; Device: The Bonfils intubation fibrescope; Device: The GlideScope Ranger; Device: The Supraglottic Airway Laryngopharyngeal Tube (SALT)
- Scenario 5: Swollen tongue (Experimental): ETI performed during mannikin swollen tongue scenario
  Interventions: Device: The Miller Laryngoscope; Device: The Bonfils intubation fibrescope; Device: The GlideScope Ranger; Device: The Supraglottic Airway Laryngopharyngeal Tube (SALT)
- Scenario 6: Immobilized cervical spine (Experimental): ETI performed during mannikin immobilized cervical spine scenario
  Interventions: Device: The Miller Laryngoscope; Device: The Bonfils intubation fibrescope; Device: The GlideScope Ranger; Device: The Supraglottic Airway Laryngopharyngeal Tube (SALT)

INTERVENTIONS:
Device: The Miller Laryngoscope — Direct laryngoscopy
Device: The Bonfils intubation fibrescope — Optical laryngoscopy
Device: The GlideScope Ranger — Videolaryngoscopy
Device: The Supraglottic Airway Laryngopharyngeal Tube (SALT) — Blind intubation

SUMMARY:
The purpose of this study was to compare the four different intubation devices in 6 different scenarios.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (paramedics, nurses, physicians)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | 1 month
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | 1 month
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
POGO score | 1 month
  self-reported percentage of glottis opening (POGO) score
VAS score | 1 month
  participants were asked which method they would prefer in a real-life resuscitation.
Cormack-Lehane grading | 1 month
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Andrzej Kurowski, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland